CLINICAL TRIAL: NCT03534648
Title: A Phase 1, Open Label, Two-cohort, Non-randomized Fixed Sequence Study To Evaluate The Pharmacokinetic Drug Drug Interaction Between Pf-05221304 And Pf-06865571 In Healthy Adult Subjects
Brief Title: Evaluation of Pharmacokinetic Drug Drug Interaction Between PF-05221304 And PF-06865571 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C3711002; DDI (Other: Alias Study Number); 2018-000694-70 (EudraCT Number)
Record Dates: First submitted 2018-04-12; First posted 2018-05-23 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Effect of PF-05221304 on PF-06865571 PK (Experimental)
  Interventions: Drug: PF-06865571 administered Day 7-14; Drug: PF-05221304 administered Day 1-14
- Effect of PF-06865571 on PF-05221304 PK (Experimental)
  Interventions: Drug: PF-06865571 administered Day 1-14; Drug: PF-05221304 administered Day 7-14

INTERVENTIONS:
Drug: PF-06865571 administered Day 7-14 — PF-06865571 administered Q12hr on Days 7-14
  Arms: Effect of PF-05221304 on PF-06865571 PK
Drug: PF-06865571 administered Day 1-14 — PF-06865571 administered Q12hr on Day 7-14
  Arms: Effect of PF-06865571 on PF-05221304 PK
Drug: PF-05221304 administered Day 1-14 — PF-05221304 administered Q12hr on Days 1-14
  Arms: Effect of PF-05221304 on PF-06865571 PK
Drug: PF-05221304 administered Day 7-14 — PF-05221304 administered Q12hr Days 7-14
  Arms: Effect of PF-06865571 on PF-05221304 PK

SUMMARY:
Drug drug interaction study between PF-05221304 and PF-06865571

DETAILED DESCRIPTION:
A Phase 1, Open Label, Two-cohort, Non-randomized Fixed Sequence Study To Evaluate The Pharmacokinetic Drug Drug Interaction Between Pf-05221304 And Pf-06865571 In Healthy Adult Subjects

ELIGIBILITY:
Inclusion criteria:

1. Healthy female subjects of nonchildbearing potential and/or male subjects.
2. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
2. Any condition possibly affecting drug absorption.
3. A positive urine drug test.
4. Screening supine BP 140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest.
5. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec.

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Arm 1: PF-05221304 Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Day 7, 0-12 hours and Day 14 0-12 hours
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 12 hours.
Arm 1: PF-05221304 Maximum observed concentration from Time Zero to End if Dosing Interval (Cmax) | Day 7, 0-12 hours and Day 14 0-12 hours
  Maximum observed concentration from Time Zero to End if Dosing Interval (Cmax)
Arm 2: PF-06865571 Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Day 7, 0-12 hours and Day 14 0-12 hours
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 12 hours.
Arm 2: PF-06865571 Maximum observed concentration from Time Zero to End if Dosing Interval (Cmax) | Day 7, 0-12 hours and Day 14 0-12 hours
  Maximum observed concentration from Time Zero to End if Dosing Interval (Cmax)

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to 28 days after last dose of study medication
  Treatment-emergent AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3711002&StudyName=A+Phase+1%2C+Open+Label%2C+Two-cohort%2C+Non-randomized+Fixed+Sequence+Study++To+Evaluate+The+Pharmacokinetic+Drug+Drug+Interaction+Between+Pf-05221304+And+Pf-06865571+In+Healthy+Adult+Subjects